CLINICAL TRIAL: NCT02835807
Title: Likes Pins and Views: Engaging Moms on Teen Indoor Tanning Thru Social Media
Brief Title: Engaging Moms on Teen Indoor Tanning Through Social Media
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klein Buendel, Inc. (Industry)
Collaborators: East Tennessee State University (Other); Colorado State University (Other); University of Connecticut (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0301; 5R01CA192652 (NIH)
Record Dates: First submitted 2016-07-14; First posted 2016-07-18 (Estimated); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Skin Cancer
Keywords: skin cancer
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Health Chat including Indoor Tanning (Experimental): Facebook group, Health Chat, which provides information via posts within the private group about a wide variety of health topics (e.g. tobacco use, body image) with 25% of all of the content being about indoor tanning. Indoor tanning-related content was developed by the investigators and a social media marketing expert using information from published literature on IT risk factors, evidence-based intervention content from published trials targeting IT reduction, public health campaigns from major non-profit organizations (e.g., CDC, Skin Cancer Foundation, etc.), and investigator-developed video-recorded interviews of local mothers and professionals about the risks of indoor tanning, experiences with skin cancer, and mother-daughter communication role modeling.
  Interventions: Behavioral: Health Chat including Indoor Tanning
- Health Chat excluding Indoor Tanning (Active Comparator): Facebook group, Health Chat, which provides information via posts within the private group about a wide variety of health topics (e.g. tobacco use, body image), but does not include any content about indoor tanning. The designated number of posts (25%) assigned to the indoor tanning content in the intervention group will be assigned to prescription drug use in the control arm. In order to keep number and frequency of posts standardized between the two groups, prescription drug use was selected to replace the indoor tanning content for the control arm.
  Interventions: Behavioral: Health Chat excluding Indoor Tanning

INTERVENTIONS:
Behavioral: Health Chat including Indoor Tanning — Participants in the intervention join a private Facebook group to participate in the Health Chat program. The group is not viewable to the public, including other Facebook users. The content of Health Chat is designed primarily for mothers, the participants in the group. Posts will occur twice daily for 12 months for a total of 720 posts. Each group will be hosted by a moderator who is responsible for managing the intervention goals and mothers' engagement. Mothers likely will not continuously engage with a social media campaign that is limited only to indoor tanning. To engage mothers in the Health Chat program, content addressing several major health and wellness topics relevant to adolescent girls and their mothers will be posted.
  Arms: Health Chat including Indoor Tanning
Behavioral: Health Chat excluding Indoor Tanning — In the comparison condition, 25% of the posts will be about prescription drug abuse and misuse. Prescription drug abuse was selected as control content because it is a) completely unrelated to tanning, and b) an emerging issue of great interest and relevance to young adults in east Tennessee. This 25% segment of posts is the only difference between the intervention and comparison conditions.
  Arms: Health Chat excluding Indoor Tanning

SUMMARY:
A sample of mothers in Tennessee are recruited to a group-randomized pretest-posttest controlled trial evaluating the effect of a social media campaign to decrease mothers' permissiveness for daughters to indoor tan. The primary outcomes is mothers' permissiveness for indoor tanning by daughters. Secondary outcomes are mother's indoor tanning prevalence and their support for stricter bans on indoor tanning by minors.

DETAILED DESCRIPTION:
Indoor tanning (IT) elevates the risk for melanoma, which is now the most common cancer in women aged 25-29. To reduce melanoma morbidity and mortality, some states have issued complete bans on IT by minors, while others require parental permission for minors to indoor tan. Unfortunately, parental consent policies have suffered from low compliance due to industry non-compliance,likely due to insufficient policy enforcement, and parents' lack of awareness of the dangers of IT. Little attention has been paid to creating health communication that maximizes the effectiveness of IT policy, including both parental consent and bans. Mothers are an important target, because their permissiveness and IT behavior are strong predictors of daughters' IT. Teen girls often initiate IT with their mothers. and further, girls who first experience IT with their mothers begin at an earlier age, become more habitual tanners, and are more resistant to change.Thus, mothers of teen girls are a significant target for interventions to reduce IT and an effective campaign for mothers has the potential to reduce the prevalence of IT in adolescent girls and the incidence of melanoma in young women. Recent research indicates that well-crafted communication can reduce maternal permissiveness but such communication has not been tested as a strategy specifically for maximizing IT policies. A campaign that aims to a) inform mothers of IT risks b) highlight how their IT permissiveness will influence their child's current and future risks,and c) provide them with effective messages to convince daughters not to indoor tan will be developed and delivered via Facebook to maximize the effectiveness of parental-permission laws, the most prevalent IT policy in the United States. The campaign will be evaluated in a group-randomized pretest-posttest controlled trial that enrolls mothers and adolescent teen daughters aged 14 to 17 years old. Participants will be randomized to receive entry into one of two private Facebook groups that will deliver health campaigns lasting one year. In the intervention group, participants will receive a health-focused feed in which 25% of posts are focused on IT. In the control condition, participants will receive the same health-focused feed but instead of 25% of posts focused on IT, 25% of posts will focus on prescription drug abuse and misuse. Randomization will occur at the level of the Facebook private groups; 30-50 mothers from the same community will participate in each Facebook private group for a total of 50 Facebook groups recruited over the trial period. Assessment points will occur at baseline and again at 6-months and 1-year post-intervention. The primary outcome will be reduction in mothers' permissiveness regarding their teen daughter's use of indoor tanning and secondary outcomes will be increase in teen daughters' perception of their mother's permissiveness,and reduction in IT by both mothers and daughters.

ELIGIBILITY:
Inclusion Criteria (Mothers):

* Live in Tennessee
* Have a daughter aged 14 to 17
* Register for the social media campaign
* Consent to participate
* Read English
* Complete the online baseline survey
* Daughter provides assent to participate
* Have a Facebook account or be willing to create one

Exclusion Criteria (Mothers):

* Not reading English
* Living outside Tennessee
* Daughter not assenting to participate

Inclusion Criteria (Daughters)

* Age 14-17
* Provide assent for mother to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1607 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Mothers' Permissiveness for Daughters to Indoor Tan | Baseline, 6-month, and 1 year follow-up
  Mothers' permissiveness for daughters to indoor tan will be assessed using 6 Likert-type items (1=strongly disagree, 5=strongly agree) assessing permissiveness toward their teenage daughter's indoor tanning. Example items include, "I would allow my daughter to indoor tan," and "I think it's OK for my daughter to indoor tan." Daughters will be asked the same 6 items to assess their perceptions of mothers' permissiveness. This measure has been used with a national teen sample. Maternal permissiveness will be assessed at baseline and both follow-ups by the combined average ratings across the six items.

SECONDARY OUTCOMES:
Change in Mothers' Indoor Tanning Prevalence | Baseline, 6-month, and 1 year follow-up
  Prevalence of indoor tanning will be assessed by asking mothers to report on their indoor tanning behavior using a single open-ended item, i.e., "How many times between December 1, 2015 and March 31, 2016 have you used a tanning bed or booth?" The December to March period was selected to control for seasonality; indoor tanning is most frequent during winter and early spring. In addition, intention to indoor tan will be assessed, i.e., How likely is it that you will indoor tan in the next 3 months/6 months/12 months (7-point Likert response scale), along with intention to get a sunless tanning treatment in the next 12 months. Indoor tanning prevalence and intentions will be assessed at baseline and both follow-ups.
Change in Daughters' Indoor Tanning Prevalence | Baseline, 6-month, and 1 year follow-up
  Prevalence of indoor tanning will be assessed by asking daughters to report on their indoor tanning behavior using a single open-ended item, i.e., "How many times between December 1, 2015 and March 31, 2016 have you used a tanning bed or booth?" The December to March period was selected to control for seasonality; indoor tanning is most frequent during winter and early spring. In addition, intention to indoor tan will be assessed, i.e., How likely is it that you will indoor tan in the next 3 months/6 months/12 months (7-point Likert response scale), along with intention to get a sunless tanning treatment in the next 12 months. Indoor tanning prevalence and intentions will be assessed at baseline and both follow-ups.
Mothers' Support for Stricter Bans on Indoor Tanning by Minors | 13-months after randomization
  Support for strengthening bans on indoor tanning (IT) by minors will be measured via the web server which will record whether mothers click on the link to "sign" the petition to strengthen the ban on indoor tanning and forward it to their legislator.

CONTACTS AND LOCATIONS:
Overall Officials: David Buller, PhD, Principal Investigator — Klein Buendel, Inc.; Sherry Pagoto, PhD, Principal Investigator — University of Connecticut
Locations (4):
- United States (4):
  - Colorado State University, Fort Collins, Colorado
  - Klein Buendel, Inc., Golden, Colorado
  - University of Connecticut, Storrs, Connecticut
  - East Tennessee State University, Johnson City, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buller D, Walkosz B, Henry K, Woodall WG, Pagoto S, Berteletti J, Kinsey A, Divito J, Baker K, Hillhouse J. Promoting Social Distancing and COVID-19 Vaccine Intentions to Mothers: Randomized Comparison of Information Sources in Social Media Messages. JMIR Infodemiology. 2022 Aug 23;2(2):e36210. doi: 10.2196/36210. eCollection 2022 Jul-Dec. PMID 36039372
- [Derived] Buller DB, Pagoto S, Henry K, Berteletti J, Walkosz BJ, Bibeau J, Baker K, Hillhouse J, Arroyo KM. Human Papillomavirus Vaccination and Social Media: Results in a Trial With Mothers of Daughters Aged 14-17. Front Digit Health. 2021 Sep 3;3:683034. doi: 10.3389/fdgth.2021.683034. eCollection 2021. PMID 34713152
- [Derived] Pagoto SL, Baker K, Griffith J, Oleski JL, Palumbo A, Walkosz BJ, Hillhouse J, Henry KL, Buller DB. Engaging Moms on Teen Indoor Tanning Through Social Media: Protocol of a Randomized Controlled Trial. JMIR Res Protoc. 2016 Nov 29;5(4):e228. doi: 10.2196/resprot.6624. PMID 27899339